CLINICAL TRIAL: NCT01867437
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Multiple Dose, 2-Period Crossover Study to Evaluate the Effect of RM-493 on Energy Expenditure in Obese Subjects
Brief Title: Effects of RM-493 on Energy Expenditure in Obese Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 130136; 13-DK-0136
Record Dates: First submitted 2013-05-22; First posted 2013-06-04 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Obesity; Morbid Obesity
Keywords: 24 Hour Energy Expenditure; Resting Energy Expenditure; Obesity; Healthy Volunteers
MeSH Terms: conditions — Obesity; Obesity, Morbid | interventions — setmelanotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RM-493 (Active Comparator): Double blind RM-493 will be administered at a dose of 1 mg/24 hrs via subcutaneous infusion for 3 days
  Interventions: Drug: RM-493
- Placebo (Placebo Comparator): Double blind placebo will be administered via subcutaneous infusion for 3 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Sterile solution (vehicle) for subcutaneous infusion
  Arms: Placebo
Drug: RM-493 — Sterile solution (2mg/ml) for subcutaneous infusion
  Arms: RM-493

SUMMARY:
Background:

- RM-493 is a drug that stimulates parts of the brain that control eating and metabolism. It has helped to reduce body weight and improve insulin sensitivity in lab tests. However, it is not fully known whether RM-493 causes weight loss by just decreasing appetite or by increasing metabolism or both. Researchers want to see how RM-493 affects metabolism and hormones that affect the metabolic rate. They also want to see how RM-493 affects appetite by assessing feelings of hunger and fullness. They will study this drug in people who are obese but are otherwise in good health.

Objectives:

- To see how RM-493 affects metabolic rate and appetite in obese but otherwise healthy individuals.

Eligibility:

- Individuals between 18 and 50 years old who are obese (body mass index between 30 and 40 kg/m2) but are otherwise healthy.

Design:

* The study consists of three phases. The first phase is the screening visit. The second phase is an 8-day inpatient stay. The final phase is a follow-up phone call one week after the end of the second phase.
* Participants will be divided into two groups. One group will receive the study drug first, followed by a placebo. The other group will receive the placebo followed by the study drug. The study drug and placebo will be given under the skin for 3 days each by a small device (OmniPod) that normally is used to give insulin to people with diabetes.
* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. They will also meet with a dietitian. The OmniPod device will be demonstrated before use.
* Participants will have the following procedures during their 8-day inpatient stay:
* Daily exercise routine (walking on treadmill) after setting a comfortable pace (miles per hour) during an exercise test
* Wear physical activity monitors
* Body composition study to measure amounts of fat and muscle
* Calorie controlled study diet
* Study drug/placebo dose through the OmniPod (Days 2 through 4 and 5 through 7)
* Metabolic rate studies using a cart or the metabolic chamber
* Daily blood samples
* Urine collection for 24 hours
* Questions about weight history and appetite
* About a week after the inpatient stay, participants will have a followup phone call to ask about any side effects from the study.

DETAILED DESCRIPTION:
Obesity is a chronic relapsing health problem and a strong risk factor for type 2 diabetes, hypertension, heart disease and stroke. Life expectancy is shorter in obese individuals who often suffer from costly related co-morbidities such as certain cancers, liver disease, osteoarthritis, sleep apnea and depression. Weight loss improves the co-morbidities. Diet and exercise are effective in the short term, but are rarely effective over a span of years. New therapies are needed especially for patients with obesity. The melanocortin system, and specifically, melanocortin 4 receptor (MC4R) is involved in the regulation of energy homeostasis and body weight. This role is validated in human genetic mutations, and in animal models of obesity, stimulation of MC4R reduces food intake and increases metabolic rate, causing a reduction in body weight.

RM-493 is a potent, selective peptide agonist for the MC4R that suppressed food intake and reduced body weight in preclinical studies. RM-493 has been studied in single dose and multiple ascending dose clinical studies in obese volunteers. This study is a randomized, double-blind, placebo-controlled, multiple-dose, 2-period, crossover study to assess the effects of RM-493 on resting energy expenditure measured in a room calorimeter. Twelve obese but otherwise healthy adult subjects between the ages of 18 and 50 inclusive, will be enrolled and randomized to one of 2 treatment sequences (RM-493 then placebo; or placebo then RM-493) over an 8-day study interval. Components of 24-hour energy expenditure, exercise induced energy expenditure, spontaneous physical activity, respiratory quotient, safety and pharmacokinetic data will be collected.

ELIGIBILITY:
* INCLUSION CRITERIA:

Male and female subjects aged 18 to 50 years at screening who meet the following inclusion and exclusion criteria will be eligible for enrollment:

* Able to provide written informed consent prior to any study procedures, and be willing and able to comply with study procedures
* Body mass index of 30-40 kg/m(2)
* Subjects who are medically healthy with normal or clinically insignificant screening results (laboratory profiles, medical histories, electrocardiograms and physical examination)
* Female subjects must have negative serum or urine pregnancy tests and must not be lactating. For females able to bear children, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control or abstinence must be used/ practiced throughout the study. Female subjects unable to bear children must have this documented in the case report form (CRF) (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]). Post-menopausal status will be confirmed by follicle stimulating hormone (FSH).
* Female subjects must have a negative serum pregnancy test prior to administering the OmniPod in both Period 1 and Period 2 to continue in the study.
* Males with female partners of childbearing potential must agree to use two medically acceptable forms of contraception as described above, with one of the two forms being condom with spermicide, from the Screening Period through the follow up phone call after completion of study treatment. Males with female partners of childbearing potential who themselves are surgically sterile (status post vasectomy) must agree to use condoms with spermicide over the same period of time.

EXCLUSION CRITERIA:

* Pregnant or lactating women
* Any clinically significant abnormalities on screening laboratories or physical examination as determined by the Investigator
* Abnormal 12-lead electrocardiogram (ECG) except minor deviations deemed to be of no clinical significance by the Investigator
* ALT or AST > 1.5 times the upper limit of normal (ULN) during screening
* Treated or untreated hypertension or blood pressure 140/90
* Treated or untreated diabetes diagnosed as fasting plasma glucose 126 or a HbA1c 6.5%
* TSH outside of the normal range
* Active or history of any significant medical condition such as and including renal, hepatic, pulmonary, gastrointestinal, cardiovascular, genitourinary, endocrine, immunologic, metabolic, neurologic or hematological disease.
* Clinical symptoms of or treatment for sleep apnea (severe snoring, excessive daytime somnolence)
* Any history of cancer, including personal history or close family history (parents or siblings) of melanoma; and/or personal history of multiple atypical nevi, nevoid basal cell carcinoma syndrome, or a personal history of non-melanoma skin cancer.
* Bariatric surgery
* History of recent surgery (within 60 days of screening)
* Current or recent (within last month) infection or viral illness
* Prescription drug use including topical steroids and inhalers, and non-prescription medicines with sympathomimetic actions (eg decongestants) if not stopped 1 week prior to and throughout the admission.
* Weight loss or gain of greater than 3% of body weight in last 3 months
* Inflexible dietary restrictions
* Actively training athletes (collegiate or professional level)
* Cigarette smoking (must be completely nonsmoking for at least 2 months)
* Dependence on caffeine, alcohol or drugs; unable or unwilling to abstain completely from caffeine and related substances for 72 hours prior to study and throughout the study
* Claustrophobia or other psychiatric conditions that would preclude participation in all aspects of the study
* Unable or unwilling to wear an insulin pump for the 6 days of treatment during the study (to deliver test drug and placebo)
* Participation in an investigational clinical study within the 30 days prior to dosing in the present study
* Any other reason, which in the opinion of the Investigator, would confound proper interpretation of the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Resting energy expenditure measured in a room calorimeter during continuous subcutaneous infusion of RM-493 or placebo in obese healthy subjects | day 4 and day 7

SECONDARY OUTCOMES:
Total energy expenditure measured in a room calorimeter during continuous subcutaneous infusion of RM-493 or placebo in obese healthy subjects | day 4 and day 7

CONTACTS AND LOCATIONS:
Overall Officials: Monica C Skarulis, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stein CJ, Colditz GA. The epidemic of obesity. J Clin Endocrinol Metab. 2004 Jun;89(6):2522-5. doi: 10.1210/jc.2004-0288. PMID 15181019
- [Background] Withrow D, Alter DA. The economic burden of obesity worldwide: a systematic review of the direct costs of obesity. Obes Rev. 2011 Feb;12(2):131-41. doi: 10.1111/j.1467-789X.2009.00712.x. PMID 20122135
- [Background] Nguyen DM, El-Serag HB. The epidemiology of obesity. Gastroenterol Clin North Am. 2010 Mar;39(1):1-7. doi: 10.1016/j.gtc.2009.12.014. PMID 20202574
- [Derived] Chen KY, Muniyappa R, Abel BS, Mullins KP, Staker P, Brychta RJ, Zhao X, Ring M, Psota TL, Cone RD, Panaro BL, Gottesdiener KM, Van der Ploeg LH, Reitman ML, Skarulis MC. RM-493, a melanocortin-4 receptor (MC4R) agonist, increases resting energy expenditure in obese individuals. J Clin Endocrinol Metab. 2015 Apr;100(4):1639-45. doi: 10.1210/jc.2014-4024. Epub 2015 Feb 12. PMID 25675384
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-DK-0136.html